CLINICAL TRIAL: NCT07082608
Title: Impact of Weight Loss From Endoscopic Sleeve Gastropathy (ESG) Plus Life Style Modification VS Life Style Modification Alone on Obstructive Sleep Apnea (OSA) Patients With Obesity - Randomized Controlled Trial
Brief Title: Effect of Weight Loss From ESG Plus Lifestyle Changes vs. Lifestyle Changes Alone in Sleep Apnea Patients
Acronym: OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Director Endoscopy (Center for Obesity and Metabolic Therapy), Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESGVSLMOS
Record Dates: First submitted 2025-07-07; First posted 2025-07-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: OSA - Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: (ESG + Lifestyle Modification) (Experimental): ESG is an endoluminal procedure similar to sleeve gastrectomy targeting the shape of the stomach. The targeted shape is a tubular gastric body with a small pouch in the fundus. The study procedure will be conducted using the Over Stitch endoscopic suturing system according to the Instructions for Use under general anesthesia.
  Participants will follow a structured program involving a low-calorie diet (typically 1200-1500 kcal/day), regular physical activity (150 minutes of moderate-intensity exercise per week), and behavioural therapy sessions.
  Interventions: Device: Endoscopic Sleeve Gastropathy; Other: Lifestyle Modification alone
- Group B: (Lifestyle Modification Alone) (Experimental): Same as described above (Group A), without the ESG procedure.
  Interventions: Other: Lifestyle Modification alone

INTERVENTIONS:
Device: Endoscopic Sleeve Gastropathy — Weight loss through diet, exercise, and behavioural changes positively impacts sleep quality. Reduction in body weight can alleviate OSA symptoms and improve overall sleep architecture1,2,3 Surgical weight loss procedures play a crucial role in managing obesity-related health issues, including OSA.4 Endobariatric procedures, including Endoscopic Sleeve Gastroplasty (ESG), have gained attention as a weight loss solution with the potential for improving obesity-related health issues.
  ESG involves suturing the stomach to reduce its size, limiting food intake. Unlike traditional bariatric surgeries, ESG doesn't require incisions. ESG has shown promise in achieving clinically significant weight loss, up to 20% of TBWL. By reducing stomach capacity, it promotes satiety and calorie restriction. ESG is generally safe, with fewer complications compared to more invasive procedures
  Arms: Group A: (ESG + Lifestyle Modification)
Other: Lifestyle Modification alone — Participants will follow a structured program involving a low-calorie diet (typically 1200-1500 kcal/day), regular physical activity (150 minutes of moderate-intensity exercise per week), and behavioural therapy sessions.

SUMMARY:
Study Overview:

Obesity and Obstructive Sleep Apnea (OSA) are strongly linked. This study aims to understand whether a procedure called Endoscopic Sleeve Gastroplasty (ESG), along with lifestyle changes like healthy eating and regular exercise, can help improve symptoms of OSA in people with obesity.

What is Obstructive Sleep Apnea (OSA)?

OSA is a condition where your breathing repeatedly stops and starts during sleep. This happens when the airway becomes blocked-often due to extra fat around the neck and throat in people with obesity. These breathing interruptions can lead to poor sleep quality, daytime tiredness, mood issues, and long-term health risks like high blood pressure and heart problems.

Why Does Weight Matter?

Obesity is a major cause of OSA. Being overweight can cause:

Narrowing of the airway

More inflammation in the body

Hormonal changes

Difficulty breathing properly during sleep

Losing weight can reduce these problems, ease OSA symptoms, and help improve sleep. Even a moderate amount of weight loss can make a big difference.

How Can People Lose Weight?

Many people try to lose weight through:

Diet changes

Exercise

Behavioural changes like mindful eating

These methods can help, but some people find it hard to lose enough weight or keep it off. That's where medical procedures like ESG can help.

What is ESG (Endoscopic Sleeve Gastroplasty)?

ESG is a non-surgical, minimally invasive weight-loss procedure. It works by reducing the size of your stomach using stitches (done through a tube inserted through your mouth-no cuts or incisions on the body). A smaller stomach means you feel full sooner and eat less.

Benefits of ESG:

Helps you lose weight (up to 20% of total body weight)

Lower risk of complications than traditional surgery

Short recovery time

No hospital stay in most cases

What Does the Research Say So Far?

Some early studies have shown that ESG can help people lose a significant amount of weight and may also improve conditions related to obesity, such as OSA.

One study followed 99 people for a year after ESG. About 30% had OSA at the start. After the procedure, many reported improvement in their OSA symptoms.

Another study compared ESG with a more invasive surgery (laparoscopic sleeve gastrectomy or LSG). While LSG led to more weight loss, both groups showed similar improvements in OSA symptoms.

This shows that ESG may be a good option for improving OSA, but more research is needed to fully understand its benefits.

Why Is This Study Important?

With obesity and OSA becoming more common, it is important to find effective and safe treatments. This study will help us learn:

How much ESG can improve sleep and breathing in people with OSA

Whether combining ESG with lifestyle changes is better than lifestyle changes alone

How ESG impacts other health problems linked to obesity

What We Hope to Learn:

We believe that weight loss from ESG will:

Reduce the severity of OSA

Improve sleep quality

Improve overall health

The results of this study could help guide future treatment options for people with obesity and sleep apnea.

DETAILED DESCRIPTION:
Obesity increases the risk of Obstructive Sleep Apnea (OSA), a condition where breathing stops during sleep. This study aims to find out whether Endoscopic Sleeve Gastroplasty (ESG) with lifestyle changes (like diet and exercise) improves OSA symptoms better than lifestyle changes alone. ESG is a non-surgical procedure that reduces stomach size to help with weight loss. Early studies show ESG can lead to weight loss and may reduce OSA symptoms, but more research is needed. This study will compare both treatment approaches to see which is more effective in improving sleep and overall health in people with obesity and OSA.

1. Primary Endpoints:

   Change in OSA severity (measured by apnea-hypopnea index, AHI) from baseline at 12 months after study procedure by group.
2. Secondary Endpoints:

   Study procedure and / or device related SAEs for the ESG group only Responders to weight loss (≥ 10% Total Body Weight Loss, TBWL) with reduction in OSA severity (AHI reduction ≥ 50%) at 12 months after study procedure by group Weight loss (TBWL%) at each study visit by group Improvement in sleep quality (assessed using validated sleep questionnaires) from baseline at 12 months after study procedure by group Epworth Sleepiness Scale (ESS) Pittsburgh Sleep Quality Index (PSQI) Change in OSA severity from baseline at 24 months after study procedure for the ESG group Responders to weight loss (≥ 10% Total Body Weight Loss, TBWL) with reduction in OSA severity (AHI reduction ≥ 50%) at 24 months after study procedure for the ESG group
3. Additional Endpoints:

Adverse event frequency related to the study procedure Responders to weight loss at each study visit by randomization group Change in OSA severity at each study visit by group Improvement in sleep quality from baseline at each study visit by group Changes in metabolic parameters: HbA1c, fasting glucose, lipid profile, and liver profile.

Changes in blood pressure and inflammatory markers (e.g., hs-CRP). Improvement in quality of life (assessed using validated questionnaires) from baseline at each study visit by group SF-36 IWQOL LITE-CT

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18years.
2. Obesity defined by ethnic specific BMI cut-offs through < 40 kg/m².
3. Diagnosed with moderate to severe OSA (Apnea-Hypopnea Index [AHI] ≥15).
4. Stable weight (< 5 kg change) within 3 months prior to screening
5. Failure or inadequate weight loss with conservative methods:

   1. lifestyle modification. and/or
   2. anti-obesity medications
6. No planned additional weight loss treatments (i.e. OTC supplements, pharmacotherapy or bariatric surgery) during the first 12-months following study treatment
7. Willingness to comply with the study protocol, including in office follow-up visits and lifestyle modifications.
8. Able to sign, understand, and sign a written Informed Consent Form to participate in the study.

Exclusion Criteria:

1. Any previous or planned surgery for sleep apnea or major ear, nose, or throat surgery
2. Significant craniofacial abnormalities that may affect breathing
3. Diagnosis of central or mixed sleep apnea, or diagnosis of Cheyne-Stokes Respiration Obesity related
4. History of disorder, other than OSA, associated with insomnia or excessive daytime sleepiness
5. Obesity induced by other endocrinologic disorders, or monogenetic or syndromic forms of obesity
6. Active device treatment of OSA other than continuous positive airway pressure therapy
7. Requires the use of supplemental oxygen
8. Previous bariatric surgery or any other gastrointestinal surgery where primary ESG will not be feasible.
9. Active inflammatory bowel disease.
10. Current or planned pregnancy or breastfeeding while participating in the study.
11. Severe cardiopulmonary conditions contraindicating endoscopy.
12. Uncontrolled psychiatric disorders.
13. Eating disorder that will impact the ability of the subject to follow the lifestyle modification program
14. History of substance abuse.
15. Use of any over-the-counter or prescription medications that could affect the evaluation of excessive sleepiness
16. Type 2 diabetics that has had a change within 3 months of the screening visit or planned change in medication for blood sugar management that has thee potential to impact weight loss (i.e. GLP-1 medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2029-05-19 (Estimated); Study Completion 2029-05-19 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Apnea Severity (AHI= Apnea Hypopnea Index) After 12 Months of Treatment: ESG Plus Lifestyle vs. Lifestyle Alone | 12 Months
  We will measure the change in Apnea-Hypopnea Index (AHI) score from baseline to 12 months after treatment, comparing the ESG + lifestyle group to the lifestyle-only group.

SECONDARY OUTCOMES:
Reduction in OSA Severity with Weight Loss | 12 months
  Percentage of participants who achieve a ≥50% reduction in AHI from baseline at 12 months post-procedure.
Weight Loss (TBWL%) | Up to 24 Months
  Total Body Weight Loss percentage (TBWL%) at each study visit, compared between groups.
Sleep Quality Assessment | 12 Months
  Improvement in sleep quality from baseline using validated questionnaires:
  * Epworth Sleepiness Scale (ESS)
  * Pittsburgh Sleep Quality Index (PSQI)
Responder Rate to Weight Loss | 12 and 24 Months
  Proportion of participants achieving ≥10% TBWL at 12 and 24 months post-procedure.
Change in OSA Severity at 24 Months in ESG Group | 24 Months
  Change in AHI from baseline to 24 months after ESG procedure.
Device- or Procedure-Related SAEs | 24 Months
  Number of Serious Adverse Events (SAEs) related to the procedure or device in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Kalapala, MD, DNB, Principal Investigator — Asian Institute of Gastroeterology
Locations (1):
- Asian Institute Of Gastroenterology Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandre F, Lapergola A, Vannucci M, Pizzicannella M, D'Urso A, Saviano A, Mutter D, Vix M, Perretta S. Endoscopic management of obesity: Impact of endoscopic sleeve gastroplasty on weight loss and co-morbidities at six months and one year. J Visc Surg. 2023 Apr;160(2S):S38-S46. doi: 10.1016/j.jviscsurg.2022.12.003. Epub 2023 Jan 30. PMID 36725451
- [Background] Hedjoudje A, Abu Dayyeh BK, Cheskin LJ, Adam A, Neto MG, Badurdeen D, Morales JG, Sartoretto A, Nava GL, Vargas E, Sui Z, Fayad L, Farha J, Khashab MA, Kalloo AN, Alqahtani AR, Thompson CC, Kumbhari V. Efficacy and Safety of Endoscopic Sleeve Gastroplasty: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2020 May;18(5):1043-1053.e4. doi: 10.1016/j.cgh.2019.08.022. Epub 2019 Aug 20. PMID 31442601
- [Background] Lopez-Nava G, Sharaiha RZ, Vargas EJ, Bazerbachi F, Manoel GN, Bautista-Castano I, Acosta A, Topazian MD, Mundi MS, Kumta N, Kahaleh M, Herr AM, Shukla A, Aronne L, Gostout CJ, Abu Dayyeh BK. Endoscopic Sleeve Gastroplasty for Obesity: a Multicenter Study of 248 Patients with 24 Months Follow-Up. Obes Surg. 2017 Oct;27(10):2649-2655. doi: 10.1007/s11695-017-2693-7. PMID 28451929
- [Background] Sharaiha RZ, Kumta NA, Saumoy M, Desai AP, Sarkisian AM, Benevenuto A, Tyberg A, Kumar R, Igel L, Verna EC, Schwartz R, Frissora C, Shukla A, Aronne LJ, Kahaleh M. Endoscopic Sleeve Gastroplasty Significantly Reduces Body Mass Index and Metabolic Complications in Obese Patients. Clin Gastroenterol Hepatol. 2017 Apr;15(4):504-510. doi: 10.1016/j.cgh.2016.12.012. Epub 2016 Dec 23. PMID 28017845
- [Background] Zhang Y, Wang W, Yang C, Shen J, Shi M, Wang B. Improvement in Nocturnal Hypoxemia in Obese Patients with Obstructive Sleep Apnea after Bariatric Surgery: a Meta-Analysis. Obes Surg. 2019 Feb;29(2):601-608. doi: 10.1007/s11695-018-3573-5. PMID 30411226
- [Background] Dombrowski SU, Knittle K, Avenell A, Araujo-Soares V, Sniehotta FF. Long term maintenance of weight loss with non-surgical interventions in obese adults: systematic review and meta-analyses of randomised controlled trials. BMJ. 2014 May 14;348:g2646. doi: 10.1136/bmj.g2646. PMID 25134100
- [Background] Malhotra A, Heilmann CR, Banerjee KK, Dunn JP, Bunck MC, Bednarik J. Weight reduction and the impact on apnea-hypopnea index: A systematic meta-analysis. Sleep Med. 2024 Sep;121:26-31. doi: 10.1016/j.sleep.2024.06.014. Epub 2024 Jun 15. PMID 38908268
- [Background] Hudgel DW, Patel SR, Ahasic AM, Bartlett SJ, Bessesen DH, Coaker MA, Fiander PM, Grunstein RR, Gurubhagavatula I, Kapur VK, Lettieri CJ, Naughton MT, Owens RL, Pepin JL, Tuomilehto H, Wilson KC; American Thoracic Society Assembly on Sleep and Respiratory Neurobiology. The Role of Weight Management in the Treatment of Adult Obstructive Sleep Apnea. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 15;198(6):e70-e87. doi: 10.1164/rccm.201807-1326ST. PMID 30215551